CLINICAL TRIAL: NCT03330535
Title: The Effect of Active Reminders on Oral Hygiene of Patients With Fixed Orthodontic Appliances With Different Time Intervals
Brief Title: The Effect of Active Reminders on Oral Hygiene in Orthodontics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Omar Alkadhi, Lecturer in Orthodontics and Clinic Director, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FRP/2018/27
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Oral Hygiene

STUDY DESIGN:
Intervention Model Description: Four groups of participants will be formulated. Each will will receive messages in different time interval starting from none, once a week, three times a week and daily.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Verbal oral hygiene instructions (Active Comparator): Participants will receive verbal oral hygiene instructions during routine orthodontic visits.
  Interventions: Behavioral: Verbal oral hygiene instructions
- Reminders once a week (Experimental): Participants will receive active reminders once a week.
  Interventions: Behavioral: Reminders once a week
- Reminders three times a week (Experimental): Participants will receive active reminders three times a week.
  Interventions: Behavioral: Reminders three times a week
- Daily reminders (Experimental): Participants will receive active reminders daily.
  Interventions: Behavioral: Daily reminders

INTERVENTIONS:
Behavioral: Reminders once a week — Participants in this group will receive active oral hygiene reminders through text messaging once a week.
  Arms: Reminders once a week
Behavioral: Verbal oral hygiene instructions — Participants in this group will receive verbal oral hygiene instructions during their regular orthodontic visits every 4 weeks.
  Arms: Verbal oral hygiene instructions
Behavioral: Reminders three times a week — Participants in this group will receive active oral hygiene reminders through text messaging three times a week.
  Arms: Reminders three times a week
Behavioral: Daily reminders — Participants in this group will receive active oral hygiene reminders through text messaging on a daily basis.
  Arms: Daily reminders

SUMMARY:
The aim of this study is to investigate the efficacy of text message active reminders at different time intervals of oral hygiene instructions in patients with orthodontic fixed appliances.

DETAILED DESCRIPTION:
Participants with orthodontic fixed appliances will be recruited from the university hospital clinics to receive text message reminders of oral hygiene. Four groups of participants will be formulated. Group 1 will be the control group and will not receive text messages. Group 2 will receive messages once a week. Group 3 will receive text message reminders 3 times a week. Group 4 will receive daily reminders. At baseline, after 4 weeks and after 8 weeks, gingival index and plaque index will be measured at each time point and then compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants were having orthodontic fixed appliance treatment.
* Participants were aged 12 years old and above, owned mobile phones and did not have mental or physical disabilities.
* Participants were willing to comply with given oral hygiene instructions.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in Plaque Index | At baseline, 4 weeks and 8 weeks
  Plaque index: 0, no plaque, 1, plaque seen on the tip of the explorer or with disclosing agent, 2. plaque seen with the naked eye, 3, abundance of plaque.
Change in gingival index | At baseline, 4 weeks and 8 weeks
  Gingival index: 0, normal gingiva, 1, mild inflammation - slight change in color, slight edema and no bleeding on probing, 2, moderate inflammation - redness, edema and glazing and bleeding on probing, 3, severe inflammation - marked redness and edema, ulceration and tendency to spontaneous bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Omar H Alkadhi, BDS,MS, Principal Investigator — Riyadh Colleges of Dentistry and Pharmacy
Locations (1):
- Riyadh Elm University, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No